CLINICAL TRIAL: NCT01597518
Title: A Multi-Center, Randomized, Placebo Controlled, Double-Blinded, Trial of Efficacy and Safety of Riluzole in Acute Spinal Cord Injury
Brief Title: Riluzole in Spinal Cord Injury Study
Acronym: RISCIS
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Enrollment challenges/ slow enrollment.
Sponsor: AOSpine North America Research Network (Network)
Collaborators: AO Foundation, AO Spine (Other); United States Department of Defense (U.S. Federal Agency); Rick Hansen Institute (Other); Christopher Reeve Paralysis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPN-12-001
Record Dates: First submitted 2012-05-10; First posted 2012-05-14 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Spinal Cord Injury
Keywords: Riluzole; spinal cord injury; treatment
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Riluzole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Riluzole (Experimental)
  Interventions: Drug: Riluzole
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Riluzole — 100mg BID first 24 hours after the injury; 50mg BID 2--14 days following the injury
  Arms: Riluzole
Drug: Placebo — Placebo 2x in first 24 hours; Placebo 2x day 2--14
  Arms: Placebo

SUMMARY:
The aim of this study is to evaluate efficacy and safety of riluzole in the treatment of patients with acute SCI. The primary objective is to evaluate the superiority of riluzole, at a dose of 2 x 100 mg the first 24 hours followed by 2 x 50 mg for the following 13 days after injury, as compared to placebo, in change between 180 days and baseline in motor outcomes as measured by International Standards for Neurological Classification of Spinal Cord Injury Examination (ISNCSCI) Motor Score, in patients with acute traumatic SCI, presenting to the hospital less than 12 hours after injury. Secondary objectives are to evaluate the effects of riluzole on overall neurologic recovery, sensory recovery, functional outcomes, quality of life outcomes, health utilities, mortality, and adverse events. The working hypothesis is that the riluzole treated subjects will experience superior motor, sensory, functional, and quality of life outcomes as compared to those receiving placebo, with an acceptable safety profile.

DETAILED DESCRIPTION:
At present there are over 1 million people living with Spinal Cord Injury (SCI) in North America alone, with annual costs for the acute treatment and chronic care of these patients totaling four billion dollars USD. The worldwide prevalence of SCI is unknown, with estimates ranging up to 250 million individuals. The incidence of SCI in developed countries has been estimated to be between 10 - 40 cases per million inhabitants. In spite of the immense impact of SCI at a personal and societal level, an effective and safe pharmacologic treatment for SCI, shown to improve neurological and functional outcomes at long-term follow-up, remains absent.

The final degree of neurological tissue destruction that occurs after traumatic SCI is a product of both primary and secondary injury mechanisms. The primary mechanical injury to the cord initiates a subsequent signaling cascade of deleterious down-stream events, known collectively as secondary injury mechanisms. These secondary injury mechanisms include ischemia, interstitial and cellular ionic imbalance, free radical formation, glutamatergic excitotoxicity, lipid peroxidation and generation of arachidonic acid metabolites. Although little can be done from a therapeutic standpoint to correct damage sustained during the primary injury, by mitigating the evolution of secondary injury events there is opportunity to preserve remnant viable neurological tissue and improve neurologic outcomes. There is convincing evidence from the preclinical realm that the pharmacologic agent riluzole attenuates certain aspects of the secondary injury cascade leading to diminished neurological tissue destruction in animal SCI models. Riluzole, a sodium channel blocking benzothiazole anticonvulsant, specifically exerts its neuroprotective effect by helping to maintain neuronal cellular ionic balance and by reducing the release of excitotoxic glutamate in the post-SCI setting. Several preclinical studies in the rodent SCI model have associated administration of riluzole with increased neural tissue preservation at the site of injury, in addition to improved behavioral outcomes, in comparison to administration of placebo or other sodium channel blocking drugs. In the clinical realm, while riluzole has not been studied extensively in the context of SCI, it has been widely used in the treatment of amyotrophic lateral sclerosis (ALS). A 2007 Cochrane review, summarizing the findings of 4 placebo-controlled randomized trials, concluded that at a dose of 100 mg daily, riluzole is safe and improves median survival by 2-3 months in patients with ALS. In regards to adverse events (AEs), riluzole was well tolerated, although treated patients were 2.6 times more likely to experience a three-fold increase in serum alanine transaminase (ALT) as compared to patients treated with placebo. However, this effect was found to be uniformly reversible with cessation of riluzole therapy and was only reported after several months of medication administration. Recently, the clinical safety and pharmacokinetic profile of riluzole have been studied in a multi-center pilot study in the context of traumatic SCI. A total of 36 patients received an oral dose of riluzole 50 mg twice daily for 2 weeks, with treatment initiated within 12 hours of injury for all patients. The 12 hour dosing window, as well as the 2 week duration of therapy, was chosen to match the period of medication administration to the known period of glutamatergic excitotoxicity after SCI (several minutes after injury until 2 weeks after injury). With the final analysis currently undergoing peer review, completion of this study has confirmed the acceptable safety profile of riluzole administration previously documented in the ALS literature, and has established the feasibility of conducting a large-scale efficacy trial investigating this therapy.

At present, there is no specific pharmacological therapy that is given uniformly to all patients with traumatic SCI. As a result, a placebo-controlled comparison group is ethical and justifiable.

The aim of the current trial is to evaluate efficacy and safety of riluzole in the treatment of patients with acute SCI.

The primary objective of the current Phase II/III trial is to evaluate the superiority of riluzole, at a dose of 2 x 100 mg the first 24 hours followed by 2 x 50 mg for the following 13 days after injury, as compared to placebo, in change between 180 days and baseline in motor outcomes as measured by International Standards for Neurological Classification of Spinal Cord Injury Examination (ISNCSCI) Motor Score, in patients with acute traumatic SCI, presenting to the hospital less than 12 hours after injury.

Secondary objectives are to evaluate the effects of riluzole on overall neurologic recovery, sensory recovery, functional outcomes, quality of life outcomes, health utilities, mortality, and adverse events. The working hypothesis is that the riluzole treated subjects will experience superior motor, sensory, functional, and quality of life outcomes as compared to those receiving placebo, with an acceptable safety profile.

ELIGIBILITY:
INCLUSION:

* Age between 18 and 75 years inclusive
* Able to cooperate in the completion of a standardized neurological examination by ISNCSCI standards (includes patients who are on a ventilator)
* Willing and able to comply with the study Protocol
* Signed Informed Consent Document (ICD) by patient, legal representative or witness
* Able to receive the Investigational Drug within 12 hours of injury
* ISNCSCI Impairment Scale Grade "A," "B" or "C" based upon first ISNCSCI evaluation after arrival to the hospital
* Neurological Level of Injury between C4-C8 based upon first ISNCSCI evaluation after arrival to the hospital
* Women of childbearing potential must have a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test or a negative urine pregnancy test

EXCLUSION:

* Injury arising from penetrating mechanism
* Significant concomitant head injury defined by a Glasgow Coma Scale score < 14 with a clinically significant abnormality on a head CT (head CT required only for patients suspected to have a brain injury at the discretion of the investigator)
* Pre-existent neurologic or mental disorder which would preclude accurate evaluation and follow-up (i.e. Alzheimer's disease, Parkinson's disease, unstable psychiatric disorder with hallucinations and/or delusions or schizophrenia)
* Previous history of spinal cord injury
* Recent history (less than 1 year) of chemical substance dependency or significant psychosocial disturbance that may impact the outcome or study participation, in the opinion of the investigator
* Is a prisoner
* Participation in a clinical trial of another Investigational Drug or Investigational Device within the past 30 days
* Hypersensitivity to riluzole or any of its components
* Neutropenia measured as absolute neutrophil count (ANC) measured in cells per microliter of blood of < 1500 at screening visit
* Creatinine level of > 1.2 milligrams (mg) per deciliter (dL) in males or > 1.1 mg per dL in females at screening visit
* Liver enzymes (ALT/SGPT or AST/SGOT) 3 times the upper limit of normal (ULN) at screening visit
* Active liver disease or clinical jaundice
* Acquired immune deficiency syndrome (AIDS) or AIDS-related complex
* Active malignancy or history of invasive malignancy within the last five years, with the exception of superficial basal cell carcinoma or squamous cell carcinoma of the skin that has been definitely treated. Patients with carcinoma in situ of the uterine cervix treated definitely more than 1 year prior to enrollment may enter the study
* Lactating at screening visit
* Subject is currently using, and will continue to use for the next 14 days any of the following medications which are classified as CYP1A2 inhibitors or inducers*:

Inhibitors:

* Ciprofloxacin
* Enoxacin
* Fluvoxamine
* Methoxsalen
* Mexiletine
* Oral contraceptives
* Phenylpropanolamine
* Thiabendazole
* Zileuton

Inducers:

* Montelukast
* Phenytoin

  * Note: no washout period required; if these medications are discontinued, subjects are eligible to be enrolled in the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2020-10-08 (Actual)

PRIMARY OUTCOMES:
Change in ISNCSCI Total Motor Score between 180 days and baseline | 180 Days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fehlings, MD, PhD, Principal Investigator — University Health Network, Toronto, Canada; Branko Kopjar, MD, PhD, Study Director — University of Washington
Locations (29):
- United States (20):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Santa Clara Valley Medical Center, San Jose, California
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Kansas University Medical Center, Kansas City, Kansas
  - University of Louisville, Louisville, Kentucky
  - Louisiana State University, Baton Rouge, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - University of Missouri, Columbia, Missouri
  - Washington University, St Louis, Missouri
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - UT Health Center, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Swedish Hospital, Seattle, Washington
  - University of Wisconsin - Madison, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (5):
  - John Hunter Hospital, Newcastle, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal Rehab, Ryde, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
- Canada (4):
  - University of British Columbia, Vancouver, British Columbia
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - University of Toronto Hospital, Toronto, Ontario

REFERENCES:
- [Background] Fehlings MG, Wilson JR, Frankowski RF, Toups EG, Aarabi B, Harrop JS, Shaffrey CI, Harkema SJ, Guest JD, Tator CH, Burau KD, Johnson MW, Grossman RG. Riluzole for the treatment of acute traumatic spinal cord injury: rationale for and design of the NACTN Phase I clinical trial. J Neurosurg Spine. 2012 Sep;17(1 Suppl):151-6. doi: 10.3171/2012.4.AOSPINE1259. PMID 22985381
- [Background] Fehlings MG, Wilson JR, O'Higgins M. Introduction: Spinal cord injury at the cutting edge of clinical translation: a focus issue collaboration between NACTN and AOSpine North America. J Neurosurg Spine. 2012 Sep;17(1 Suppl):1-3. doi: 10.3171/2012.6.AOSPINE12632. No abstract available. PMID 22985363
- [Background] Wilson JR, Forgione N, Fehlings MG. Emerging therapies for acute traumatic spinal cord injury. CMAJ. 2013 Apr 2;185(6):485-92. doi: 10.1503/cmaj.121206. Epub 2012 Dec 10. No abstract available. PMID 23228995
- [Background] Grossman RG, Fehlings MG, Frankowski RF, Burau KD, Chow DS, Tator C, Teng A, Toups EG, Harrop JS, Aarabi B, Shaffrey CI, Johnson MM, Harkema SJ, Boakye M, Guest JD, Wilson JR. A prospective, multicenter, phase I matched-comparison group trial of safety, pharmacokinetics, and preliminary efficacy of riluzole in patients with traumatic spinal cord injury. J Neurotrauma. 2014 Feb 1;31(3):239-55. doi: 10.1089/neu.2013.2969. Epub 2013 Oct 11. PMID 23859435
- [Background] Nagoshi N, Fehlings MG. Investigational drugs for the treatment of spinal cord injury: review of preclinical studies and evaluation of clinical trials from Phase I to II. Expert Opin Investig Drugs. 2015 May;24(5):645-58. doi: 10.1517/13543784.2015.1009629. Epub 2015 Feb 3. PMID 25645889
- [Background] Nagoshi N, Nakashima H, Fehlings MG. Riluzole as a neuroprotective drug for spinal cord injury: from bench to bedside. Molecules. 2015 Apr 29;20(5):7775-89. doi: 10.3390/molecules20057775. PMID 25939067
- [Background] Fehlings MG, Nakashima H, Nagoshi N, Chow DS, Grossman RG, Kopjar B. Rationale, design and critical end points for the Riluzole in Acute Spinal Cord Injury Study (RISCIS): a randomized, double-blinded, placebo-controlled parallel multi-center trial. Spinal Cord. 2016 Jan;54(1):8-15. doi: 10.1038/sc.2015.95. Epub 2015 Jun 23. PMID 26099215
- [Result] Chow DS, Teng Y, Toups EG, Aarabi B, Harrop JS, Shaffrey CI, Johnson MM, Boakye M, Frankowski RF, Fehlings MG, Grossman RG. Pharmacology of riluzole in acute spinal cord injury. J Neurosurg Spine. 2012 Sep;17(1 Suppl):129-40. doi: 10.3171/2012.5.AOSPINE12112. PMID 22985379
- [Result] Wilson JR, Fehlings MG. Riluzole for acute traumatic spinal cord injury: a promising neuroprotective treatment strategy. World Neurosurg. 2014 May-Jun;81(5-6):825-9. doi: 10.1016/j.wneu.2013.01.001. Epub 2013 Jan 4. PMID 23295632
- [Derived] Carroll AH, Fakhre E, Quinonez A, Tannous O, Mesfin A. An Update on Spinal Cord Injury and Current Management. JBJS Rev. 2024 Oct 24;12(10). doi: 10.2106/JBJS.RVW.24.00124. eCollection 2024 Oct 1. PMID 39446982
- [Derived] Fehlings MG, Moghaddamjou A, Harrop JS, Stanford R, Ball J, Aarabi B, Freeman BJC, Arnold PM, Guest JD, Kurpad SN, Schuster JM, Nassr A, Schmitt KM, Wilson JR, Brodke DS, Ahmad FU, Yee A, Ray WZ, Brooks NP, Wilson J, Chow DS, Toups EG, Kopjar B. Safety and Efficacy of Riluzole in Acute Spinal Cord Injury Study (RISCIS): A Multi-Center, Randomized, Placebo-Controlled, Double-Blinded Trial. J Neurotrauma. 2023 Sep;40(17-18):1878-1888. doi: 10.1089/neu.2023.0163. Epub 2023 Jul 13. PMID 37279301
- [Derived] Chow DS, Nguyen A, Park J, Wu L, Toups EG, Harrop JS, Guest JD, Schmitt KM, Aarabi B, Fehlings MG, Boakye M, Grossman RG. Riluzole in Spinal Cord Injury Study (RISCIS)-Pharmacokinetic (PK) Sub-Study: An Analysis of Pharmacokinetics, Pharmacodynamics, and Impact on Axonal Degradation of Riluzole in Patients With Traumatic Cervical Spinal Cord Injury Enrolled in the RISCIS Phase III Randomized Controlled Trial. J Neurotrauma. 2023 Sep;40(17-18):1889-1906. doi: 10.1089/neu.2022.0499. PMID 37130044
- [Derived] Satkunendrarajah K, Nassiri F, Karadimas SK, Lip A, Yao G, Fehlings MG. Riluzole promotes motor and respiratory recovery associated with enhanced neuronal survival and function following high cervical spinal hemisection. Exp Neurol. 2016 Feb;276:59-71. doi: 10.1016/j.expneurol.2015.09.011. Epub 2015 Sep 21. PMID 26394202
- See also: AOSpine North America is a non for profit foundation for excellence in spine — http://www.aospine.org